CLINICAL TRIAL: NCT03128944
Title: Development of the Blood Pressure Imager
Brief Title: Feasibility Assessment of the Blood Pressure Imager, a Continuous Blood Pressure Monitor
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Mohan Thanikachalam, Research Assistant Professor, Tufts University
Other Study IDs: 12351
Record Dates: First submitted 2017-04-21; First posted 2017-04-25 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are developing Blood Pressure Imager (BPI), which is a new technology that does not require cuffs or expensive equipment, and can be used by untrained individuals in underserved, low-resource environments at their own homes or regional care settings. Over the last one-year the investigators have developed the BPI prototype, which is ready for testing. BPI is a wrist device that includes a camera, color lights and soft membrane with a reflective coating. In this device feasibility study, the BPI will be placed over the radial artery at the wrist with the help of a wrist strap. The primary purpose of this feasibility study is to compare the BPI with a commercially available cuff-based blood pressure measuring devices.

DETAILED DESCRIPTION:
If the participant volunteers to participate in this study, after signing the informed consent, responses to background data - age, gender, height, weight, wrist circumference of dominant arm, history of high blood pressure, diabetes, high cholesterol and cardiovascular disease - will be collected; The BPI will be strapped to the right or left wrist making sure it is comfortable to the participant and the readings from the BPI will be recorded in a computer. The continuous BPI readings will be recorded for 2 minutes. Simultaneously, blood pressure readings will be obtained from a cuff-based, commercially available blood pressure measuring device placed in the same arm. The research team will take a minimum 3 and maximum 6 sets of readings. At the end of the BPI readings, we will place an ultrasound probe of the wrist at the level of the wrist to assess the size of the radial artery and depth of the artery from the skin.

Participant Timeline: The collection of the background data will take 5 to 10 mins. The placement of the BPI and cuff-blood pressure device and the data collection will take about 15 to 20 mins. The ultrasound image collection will 10 to 15 mins. Overall, the study procedures will be less than an hour.

ELIGIBILITY:
Inclusion Criteria:

* Tests will be performed with any adult volunteer who is physically and mentally able to perform the experimental tasks.

Exclusion Criteria:

* We will restrict the experiments to adult volunteers who are physically and mentally able to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study accepts adult (age of 18 years and above) volunteers with or without high blood pressure who are physically and mentally able to consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Comparison of BPI measurements with reference blood pressure measurements | 1 hour
  Comparison of BPI measurements with reference blood pressure measurements with commercially available cuff-based blood pressure measuring device

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Thanikachalam, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No